CLINICAL TRIAL: NCT05377970
Title: Implementation of a Prehabilitation Pilot Program for Individuals With Frailty Undergoing Oncologic Surgery
Brief Title: Implementation of a Prehabilitation Program for Surgical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MaineHealth (Other)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Laura Nicolais, Timothy Fitzgerald: Associate Medical Director. Oncology, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1855206
Record Dates: First submitted 2022-04-08; First posted 2022-05-17 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Prehabilitation; Oncology; Surgical Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation Intervention Program (Experimental): Patients enrolled in this arm will receive the preabilitation intervention program prior to their surgery to complete
  Interventions: Other: Thinkific Prehabilitation Exercise Program

INTERVENTIONS:
Other: Thinkific Prehabilitation Exercise Program — Prehabilitation exercise program through the Thinkific platform

SUMMARY:
Frailty is a state of increased vulnerability to stressors with increased rates of poor outcomes. Surgery is one of these stressors, and previous research has therefore shown increased rates of morbidity and mortality in frail patients undergoing surgery. Prehabilitation programs can help mitigate the negative outcomes associated with frailty. The investigators hope to implement a newly developed prehabilitation pilot program in the Maine Medical Center Surgical Oncology Clinic to initially evaluate adherence, self-efficacy, and health-related quality of life.

DETAILED DESCRIPTION:
Frailty is a state of increased vulnerability to stressors with increased rates of poor outcomes. Surgery is one of these stressors, and previous research has therefore shown increased rates of morbidity and mortality in frail patients undergoing surgery. Prehabilitation programs can help mitigate the negative outcomes associated with frailty. The investigators hope to implement a newly developed prehabilitation pilot program in the Maine Medical Center Surgical Oncology Clinic to initially evaluate adherence, self-efficacy, and health-related quality of life.

The investigators now hope to implement this prehabilitation program in the clinics at Maine Medical Center. Our long term goal is the introduce this program in all surgical specialties; but first, the investigators plan to assess adherence, patient self-efficacy, frailty and health-related quality of life through a pilot study in the surgical oncology clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years old
2. Evaluated at Maine Medical Center by surgical oncology service
3. Planned surgical intervention for gastrointestinal oncologic condition
4. Score ≥40 on Risk Analysis Index frailty screening
5. Physically able to participate in prehabilitation exercises
6. Home internet access and established email account
7. Able to understand the English language

Exclusion Criteria:

1. Patients unable to participate in exercises included in prehabilitation program
2. Patients with impaired decision making capacity
3. Those in a high risk community: prisoners and pregnant women
4. Those who do not meet the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Participant adherence to prehab program | Through study completion, on average 3 months
  Evaluate adherence through analysis of patient maintained exercise logs via number of days completed
Correlation between patient pre-program self-efficacy evaluation and measured adherence to study prehabilitation program | Through study completion, on average 3 months
  Assess self-efficacy by evaluating the relationship between pre-program Self-Efficacy for Home Exercise Program Scale (0-72) score and adherence.
Patient Satisfaction | Last day of prehabilitation program (within week prior to surgery)
  Assess patient satisfaction and barriers to adherence through a post prehab program survey.
Quality of Life (Short Form- 36 Survey) | Completed at Day 0, Two weeks, Four weeks and Last day of prehabilitation program (within week prior to surgery)
  Evaluate change in health-related quality of life before and after participation in the prehabilitation program.
Frailty (Risk Analysis Index) | Evaluated on Day 0 and at last visit prior to surgery, an average of 3 months
  Evaluate change in frailty using Risk Analysis Index before and after participation in the prehabilitation program.

CONTACTS AND LOCATIONS:
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT05377970/Prot_SAP_000.pdf